CLINICAL TRIAL: NCT07068191
Title: Randomized Comparative Clinical Study of the Dietary Supplement "Gepaktiv" (International Name: Phenomenon) in Comparison With Ursodeoxycholic Acid (UDCA) and Ademetionine in Patients With Metabolic Associated Fatty Liver Disease (MAFLD) and Hepatomegaly
Brief Title: Gepaktiv vs UDCA and Ademetionine in MAFLD With Hepatomegaly
Acronym: HEPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phenomen Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEP-2025-01
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-associated Fatty Liver Disease (MAFLD); Hepatomegaly; Nonalcoholic Fatty Liver (NAFL); Nonalcoholic Fatty Liver Disease (NAFLD); Fatty Liver; Fatty Liver, Alcoholic; Fatty Liver, Nonalcoholic; Fatty Liver Disease
Keywords: Hepatomegaly; Gepaktiv; Metabolic dysfunction-associated fatty liver disease (MAFLD); metabolic dysfunction-associated steatotic liver disease (MASLD); Nonalcoholic fatty liver disease (NAFLD); liver diseases; Nonalcoholic fatty liver (NAFL); Liver; Liver steatosis; Dietary supplements; Fatty Liver
MeSH Terms: conditions — Hepatomegaly; Non-alcoholic Fatty Liver Disease; Fatty Liver; Fatty Liver, Alcoholic; Liver Diseases | interventions — Ursodeoxycholic Acid; S-Adenosylmethionine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned (1:1:1) to three parallel groups for 15 days:
  1. Gepaktiv (dietary supplement, 2 capsules × 3 times/day),
  2. UDCA (10-15 mg/kg/day),
  3. Ademetionine (800-1600 mg/day). Gepaktiv is a dietary supplement; comparator arms receive standard therapy according to national guidelines.
  UDCA and Ademetionine are included as standard-of-care active comparators (not investigational drugs).
  Post-treatment follow-up is optional (up to 60 days). Blinded assessors evaluate outcomes.
Who Masked: Outcomes Assessor
Masking Description: Biochemical and imaging data are evaluated by independent assessors blinded to group assignment. Outcome assessors do not have access to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 2 (n=30) (Active Comparator): Group 2 (n=30): UDCA 10-15 mg/kg/day;
  Interventions: Drug: UDCA (Ursodeoxycholic acid)
- Group 3 (n=30) (Active Comparator): Group 3 (n=30): Ademetionine 800-1600 mg/day.
  Interventions: Drug: Ademetionine
- Group 1 (n=30) (Experimental): Participants receive dietary supplement 'Gepaktiv' (2 capsules × 3 times/day, 60 minutes before meals
  Interventions: Combination Product: Dietary supplement "Gepaktiv"

INTERVENTIONS:
Combination Product: Dietary supplement "Gepaktiv" — Dietary supplement "Gepaktiv" 60 minutes before meals 2 capsules × 3 times/day
  Arms: Group 1 (n=30)
Drug: UDCA (Ursodeoxycholic acid) — UDCA 10-15 mg/kg/day
  Arms: Group 2 (n=30)
Drug: Ademetionine — Ademetionine 800-1600 mg/day.
  Arms: Group 3 (n=30)

SUMMARY:
This study compares the effectiveness of the dietary supplement Gepaktiv with standard medications (UDCA and Ademetionine) in patients with fatty liver disease (MAFLD) and liver enlargement (hepatomegaly).

Key points:

* Participants will receive either Gepaktiv, UDCA, or Ademetionine for 15 days
* Doctors will monitor liver health through blood tests and ultrasound scans
* The study will check if Gepaktiv helps improve liver function as effectively as standard treatments.

Main measurements:

* Changes in liver enzyme levels (ALT, AST)
* Reduction in liver size
* Improvement in fat accumulation (steatosis) measured by FibroScan This research may provide evidence for a new natural option to support liver health.Data analysis will be done by an independent biostatistics

DETAILED DESCRIPTION:
This randomized, open-label, parallel-group study evaluates the hepatoprotective effects of the dietary supplement Gepaktiv (250 mg capsules) compared to ursodeoxycholic acid (UDCA) and ademetionine in 90 patients with metabolic-associated fatty liver disease (MAFLD) and hepatomegaly.

Study Design:

* Duration: 15-day treatment with optional 60-day follow-up
* 3 treatment arms (n=30 each):

  1. Gepaktiv (2 capsules × 3 times daily)
  2. UDCA (10-15 mg/kg/day)
  3. Ademetionine (800-1600 mg/day)
* Randomization: 1:1:1 block randomization

Primary Endpoints:

1. ≥30% reduction in ALT levels
2. Liver size reduction (ultrasound)
3. Improvement in FibroScan parameters (CAP for steatosis, kPa for fibrosis)

Secondary Endpoints:

* Changes in other liver enzymes (AST, GGT, bilirubin)
* Lipid profile (triglycerides, cholesterol)
* Albumin and total protein levels
* Quality of life assessment (CLDQ questionnaire)

Methodology Highlights:

* Standardized ultrasound protocol (single operator)
* Central laboratory analysis of biomarkers
* All efficacy-related assessments (FibroScan, ultrasound, and laboratory blood tests) are performed by blinded evaluators who are not involved in patient management or aware of group assignment
* Daily compliance monitoring through patient diaries

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Confirmed diagnosis of metabolic-associated fatty liver disease (MAFLD)
* Hepatomegaly confirmed by ultrasound (≥3 cm craniocaudal liver enlargement)
* ALT level between 90-150 U/L
* Steatosis ≥260 dB/m by FibroScan (CAP)
* Fibrosis ≥11 kPa by transient elastography (FibroScan)
* Ability to comply with study procedures
* Signed informed consent

Exclusion Criteria:

* Liver cirrhosis or hepatocellular carcinoma
* Pregnancy or lactation
* Known allergy to any of the study medications or supplement components
* Gallstones or biliary obstruction
* Shrunken liver on imaging
* Hepatic cysts (simple liver cysts/biliary cysts)
* Liver nodules (focal liver lesions)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in ALT levels by ≥30% from baseline | 15 days (+ optional post-observation up to 60 days).
  Proportion of participants achieving ≥30% decrease in serum ALT after 15 days of treatment
Change in liver size (ultrasound) | 15 days (+ optional post-observation up to 60 days).
  Reduction in liver enlargement (≥1 cm) measured by standardized ultrasound
Improvement in steatosis/fibrosis (FibroScan) | 15 days (+ optional post-observation up to 60 days).
  Change in CAP (steatosis) and kPa (fibrosis) scores from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Tyumen State Medical University, Tyumen, Tyumen Oblast, Russia